CLINICAL TRIAL: NCT02257957
Title: Platelet -Rich Plasma (PRP) Injection for the Treatment of Severe Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: plasmadry10
Record Dates: First submitted 2014-09-24; First posted 2014-10-07 (Estimated); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye; Sjogren Syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet -Rich Plasma (PRP) (Experimental): 15 patients with diagnosis of severe dry eye will receive PRP injection at day 0, 30,60 and 90
  Interventions: Drug: PRP injection
- Standard Care (Active Comparator): 15 patients with diagnosis of severe dry eye will receive standard of care treatment and will be revised at day 0, 30,60,90
  Interventions: Drug: Standard care Hyaluronic acid eye drops

INTERVENTIONS:
Drug: PRP injection
  Arms: Platelet -Rich Plasma (PRP)
Drug: Standard care Hyaluronic acid eye drops — : 15 patients with diagnosis of severe dry eye will receive standard of care treatment ( Hyaluronic acid eye drops 5 times per day). Objective measurements as corneal staining, Shirmer , BUT, and VA, will be determinate as subjective measurements as OSDI and treatment compliance will be evaluated at day 0-30,60 and 90
  Arms: Standard Care

SUMMARY:
Dry eye is a chronic condition that decreases function and affect visual function with severe discapacity until now treatments are based in artificial eye drops. Platelet rich plasma has emerged as a strategy for cellular restoration, the purpose of this study is to evaluate their effects in lacrimal production and safety of this intervention in patients with severe dry eye.

DETAILED DESCRIPTION:
Dry eye is a chronic condition that decreases function and affect visual function with severe discapacity until now treatments are based in artificial eye drops. Platelet rich plasma has emerged as a strategy for cellular restoration, the purpose of this study is to evaluate their effects in lacrimal production and safety of this intervention in patients with severe dry eye.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with symptomatic Dry eye

  * Shirmer ≤10 mm in 5 min
  * BUT ≤10 seconds
  * Corneal staining ≥3
  * Age range: 18 years and older.
  * Both genders and all ethnic groups comparable with the local community.
  * Able to understand and willing to sign a written informed consent
  * Able and willing to cooperate with the investigational plan.
  * Able and willing to complete all mandatory follow-up visits.

Exclusion Criteria:

* • Patients who are currently engaged in another clinical trial, unwilling or unable to give consent, to accept randomization, or to return for scheduled visits.

  * Children under 18.
  * Pregnant women or expecting to be pregnant during the study.
  * Systemic immune deficient conditions such as AIDS or under systemic immunosuppressant.
  * Concomitant use of systemic antibiotics or steroids.
  * Contact lens wear
  * Active ocular infection or allergy
  * Unable to close eyes or uncontrolled blinking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-04-20 (Actual)

REFERENCES:
- [Derived] Avila MY, Igua AM, Mora AM. Randomised, prospective clinical trial of platelet-rich plasma injection in the management of severe dry eye. Br J Ophthalmol. 2018 Jul 3:bjophthalmol-2018-312072. doi: 10.1136/bjophthalmol-2018-312072. Online ahead of print. PMID 29970389

RESULTS

PARTICIPANT FLOW:
Groups:
- Platelet -Rich Plasma (PRP): 15 patients with diagnosis of severe dry eye will receive PRP injection at day 0, 30,60 and 90
  PRP injection
Period: Overall Study
Arm/Group | Platelet -Rich Plasma (PRP) | Standard Care
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet -Rich Plasma (PRP) | Standard Care | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (3.5) | 52.7 (3.5) | 52.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Staining
Description: Surface damage to the exposed eye, assessed by staining, is graded against standard charts. According to the Oxford grade panel (Oxford Scale), the staining was graded and was classified from grade 0 to grade V (0 to 5 score). The minimum value of this scale was 0, which indicating absent surface damage, and the maximum value was 5, which meaning severe surface damages.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet -Rich Plasma (PRP) | Standard Care
Number analyzed (Participants) | 15 | 15
score on a scale | 1.2 (0.18) | 2.4 (0.18)

2. Primary Outcome: Change From Baseline in Shirmer Test
Description: The Schirmer test I (performed without anaesthesia) was completed before any drops were instilled in the eye. Standardised Schirmer strips (Biotech Vision Care, Gandhinagar, India) were bent at the notch and placed carefully over the lower lid margin as far as possible towards the temporal angle of the lids. The patient was instructed to keep his/her eyelids closed during the test. The strips remained in place for 5 min. After 5 min, the amount of moisture in each strip was measured using a millimetre scale
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Platelet -Rich Plasma (PRP) | Standard Care
Number analyzed (Participants) | 15 | 15
mm | 9.2 (1) | 5.3 (0.7)

3. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI)
Description: The OSDI consists of 12 questions on items related to the assessment of symptoms, functional limitations and environmental factors related to dry eye. It is graded on a scale of 0-4, with 0 indicating none of the time, 1 for some of the time, 2 for half of the time, 3 for most of the time and 4 indicating all the time. This is a valid and reliable instrument for measuring the severity of dry eye.
  The total OSDI score was then calculated by the following formula: OSDI = (sum of scores for all questions answered) × 100/(total number of questions answered) × 4). A score of 0-100 was obtained, related to the extent of dry eye, which a higher score representing greater symptoms severity.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet -Rich Plasma (PRP) | Standard Care
Number analyzed (Participants) | 15 | 15
score on a scale | 34 (4) | 55 (2.5)

ADVERSE EVENTS:
Arm/Group | Platelet -Rich Plasma (PRP) | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes